CLINICAL TRIAL: NCT02753140
Title: Concurrent Chemoradiotherapy in Locally Advanced Squamous Cell Carcinoma of the Head and Neck Versus Concomitant Cetuximab With Radiotherapy After Neoadjuvant Chemotherapy: a Randomized, Opened, Multicenter Phase II Trial
Brief Title: Concurrent Chemoradiotherapy(CRT) in Locally Advanced(LA) SCCHN vs Cetuximab With Radiotherapy (RT) After Neoadjuvant Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhen-zhou Yang, Director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YangZZ-2016
Record Dates: First submitted 2016-04-18; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Radiation; Docetaxel; Cisplatin

ARMS (2):
- RT concurrent with cetuximab (Experimental): Selected 60 patients with locally advanced squamous cell carcinoma of the head and neck. They will be randomized to concurrent chemoradiotherapy versus concomitant cetuximab with radiotherapy after neoadjuvant chemotherapy.To observe the curative effect of the treatment of the cetuximab
  Interventions: Drug: Cetuximab; Radiation: radiation
- RT concurrent with TP (Experimental): Selected 60 patients with locally advanced squamous cell carcinoma of the head and neck. They will be randomized to concurrent chemoradiotherapy versus concomitant cetuximab with radiotherapy after neoadjuvant chemotherapy. To observe the curative effect of concurrent radiotherapy and chemotherapy
  Interventions: Radiation: radiation; Drug: Docetaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Cetuximab
  Arms: RT concurrent with cetuximab
Radiation: radiation
Drug: Docetaxel
  Arms: RT concurrent with TP
Drug: Cisplatin
  Arms: RT concurrent with TP

SUMMARY:
Verify the effect and the incidence of oral mucositis of concurrent chemoradiotherapy in locally advanced squamous cell carcinoma of the head and neck versus concomitant cetuximab with radiotherapy after neoadjuvant chemotherapy.

The predictive effect of Apurinic/apyrimidinic endonuclease 1(APE1)/ Ref-1 protein and Apurinic/apyrimidinic endonuclease 1(APE1)/Ref-1 antibody on oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed first diagnosis of locally advanced squamous cell carcinoma of the head and neck
2. Imaging (MRI, CT, bone scan) stage Ⅲ、Ⅳa (T1-2N2M0、T3N0-2M0、T4N0-2M0) (2010AJCC staging criteria)
3. 18 years of age or older
4. Presence of at least 1 measurable lesion according to RECIST version1.1
5. DON'T accept surgery, chemotherapy or irradiation before trial entry
6. Eastern Cooperative Oncology Group(ECOG) 0 or 1
7. Expected survival period over 6months
8. Before RT randomization, bone marrow and liver and kidney function in patients with meet the following criteria:

   * Hemoglobin(HB) ≥ 100g/L, neutrophil ≥ 2.0 × 109/L and platelet ≥ 100 × 109/L
   * Total bilirubin ≤ 1.5 times the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 times the upper limit of normal;
   * More than 1.5 times the upper limit of normal serum creatinine or creatinine clearance rate ≥ 60 ml/min, urea N ≤ 200mg/L;
   * The blood glucose level: good blood glucose control, fasting glucose, 3.9-7.2mmol/L postprandial blood glucose less than 10.0mmol/L, HbA1c < 7%;
9. Signed written informed consent before any trail-related activities are carried out.

Exclusion Criteria:

1. Patients accepted chemotherapy、radiotherapy or surgery;
2. Distant metastasis before trail entry
3. Female subjects who are pregnant or breast feeding;
4. oral mucositis or oral mucositis has repeatedly made (1 times / month or more)before Chemotherapy or radiotherapy ;
5. With teeth periodontitis;
6. Any investigational medication within 30 days before trial entry;
7. Elderly patients with dry stomatitis;
8. Any unstable system diseases: including active infection, uncontrolled hypertension, unstable angina pectoris, within the last 3 months of the onset of angina, congestive heart failure, the group in June before the myocardial infarction, need serious mental disorder drug treatment, liver, kidney or metabolic diseases; mental / spiritual diseases such as Alzheimer's disease;
9. Total bilirubin > 1.5 times the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2.5 times the upper limit of normal;
10. On gastrointestinal physiology is not perfect, or absorb the obstacle syndrome, or unable to tolerate oral medication, or active peptic ulcer；
11. Past or current history of neoplasm oher than squamous cell carcinoma of the head and neck;
12. Judgment according to the researchers, there are serious harm to patient safety or affect the patients completed the study with the disease, and patient compliance with the difference;
13. known human immunodeficiency virus (HIV) infection;
14. With immunodeficiency disease, or suffer from other acquired, congenital immunodeficiency disease, or a history of organ transplantation;
15. Any disease, metabolic disorders, or physical examination or laboratory suspicion or treatment of complications in patients at high risk of drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-03 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 13 months
incidence of oral mucositis | 3 months

SECONDARY OUTCOMES:
Overall survival | 5 years
Overall response rate after induction chemotherapy | 1 month